CLINICAL TRIAL: NCT00476554
Title: A Randomized Phase II Study of Oral Sapacitabine in Patients With Advanced Cutaneous T-cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual and financial resource limitation
Sponsor: Cyclacel Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYC682-06-05; NCT00475995 (obsolete NCT alias)
Record Dates: First submitted 2007-05-19; First posted 2007-05-22 (Estimated); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Cutaneous T-cell Lymphoma (CTCL)
Keywords: CTCL
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous | interventions — sapacitabine

ARMS (2):
- Arm A: High dose (Experimental): High-dose (Arm A): 200 mg b.i.d. x 3 consecutive days per week for 2 weeks followed by 1-week rest
  Interventions: Drug: Sapacitabine
- Arm B: High dose (Experimental): Low-dose (Arm B): 100 mg b.i.d. x 3 consecutive days per week for 2 weeks followed by 1-week rest
  Interventions: Drug: Sapacitabine

INTERVENTIONS:
Drug: Sapacitabine — Sapacitabine
  Other Names: CYC682

SUMMARY:
This is an open label, randomized phase II study designed to evaluate the tolerability and response rate of high-dose and low-dose regimens in patients with advanced cutaneous T-cell lymphoma (CTCL).

DETAILED DESCRIPTION:
This is an open label, randomized phase II study designed to evaluate the tolerability and response rate of high-dose and low-dose regimens in patients with advanced cutaneous T-cell lymphoma (CTCL) who have had progressive, recurrent, or persistent disease on or following 2 systemic therapies.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with advanced CTCL
* Have had at least 2 systemic therapies
* Must have evaluable disease
* Eastern Cooperative Oncology Group performance status 0-2
* Adequate bone marrow, hepatic and renal function
* At least 3 weeks from prior therapies
* Not receiving topical steroids or have been on a stable dose of topical steroids for at least 2 weeks
* Able to swallow capsules
* At least 3 weeks from major surgery
* Agree to practice effective contraception
* Able to understand and willing to sign the informed consent form

Exclusion Criteria:

* Receiving systemic steroids
* Receiving topical or systemic retinoids or vitamin A
* Receiving radiotherapy, biological therapy,or any other investigational agents
* Uncontrolled intercurrent illness
* Pregnant or lactating women
* Known to be HIV-positive
* Active hepatitis B and/or hepatitis C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-04; Primary Completion 2012-03-01 (Actual); Study Completion 2012-03-01 (Actual)

PRIMARY OUTCOMES:
response rate in overall skin disease | over the course of study
  Decrease of lesion from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Judy H Chiao, M.D., Study Director — Cyclacel Pharmaceuticals, Inc.
Locations (3):
- United States (3):
  - Stanford University Hospitals and Clinics, Stanford, California
  - Timothy Kuzel, M.D., Chicago, Illinois
  - The University of Texas MD Anderson Cancer Center, Houston, Texas